CLINICAL TRIAL: NCT01256684
Title: DHEA Against Vaginal Atrophy (Placebo-controlled, Double-blind and Randomized Phase III Study of 3-month Intravaginal DHEA)
Brief Title: DHEA Against Vaginal Atrophy - 3-Month Efficacy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EndoCeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-231
Record Dates: First submitted 2010-12-03; First posted 2010-12-08 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Vaginal Atrophy
Keywords: Vulvar/vaginal atrophy; Atrophic Vaginitis; Dehydroepiandrosterone; DHEA; Prasterone; Vaginorm; Menopause; Intrarosa
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 0.25% DHEA (Experimental)
  Interventions: Drug: DHEA
- 0.5% DHEA (Experimental)
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: Placebo — Placebo vaginal suppository
  Arms: Placebo
Drug: DHEA — Vaginal suppository containing 0.25% (3.25 mg) DHEA; daily dosing with one suppository for 12 weeks.
  Other Names: Prasterone, Dehydroepiandrosterone
  Arms: 0.25% DHEA
Drug: DHEA — Vaginal suppository containing 0.50% (6.5 mg) DHEA; daily dosing with one suppository for 12 weeks.
  Other Names: Prasterone, Dehydroepiandrosterone
  Arms: 0.5% DHEA

SUMMARY:
The purpose of this Phase III trial is to confirm the efficacy of intravaginal dehydroepiandrosterone (DHEA) in postmenopausal women with vaginal atrophy.

ELIGIBILITY:
Main Inclusion Criteria:

* Postmenopausal women (hysterectomized or non-hysterectomized)
* Women between 40 and 75 years of age.
* Willing to participate in the study and sign an informed consent.
* Women who have self-identified symptom(s)of vaginal atrophy.
* For non-hysterectomized women, willing to have endometrial biopsy at screening and end of study.

Main Exclusion Criteria:

* Undiagnosed abnormal genital bleeding.
* Hypertension equal to or above 140/90 mm Hg.
* The administration of any investigational drug within 30 days of screening visit.
* Endometrial hyperplasia, cancer or endometrial histology showing proliferative, secretory or menstrual type characteristics at histologic evaluation of endometrial biopsy performed at screening.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Archer, MD, Principal Investigator — Clinical Research Center, Eastern Virginia Medical School, Norfolk, VA
Locations (33):
- United States (24):
  - EndoCeutics site # 39, Montgomery, Alabama
  - EndoCeutics site # 14, Tucson, Arizona
  - EndoCeutics site # 21, Sacramento, California
  - EndoCeutics site # 30, San Diego, California
  - EndoCeutics site # 17, San Diego, California
  - EndoCeutics site # 36, Denver, Colorado
  - EndoCeutics site # 42, Milford, Connecticut
  - EndoCeutics site # 45, Boynton Beach, Florida
  - EndoCeutics site # 26, Jacksonville, Florida
  - EndoCeutics site # 23, Sandy Springs, Georgia
  - EndoCeutics site # 10, Meridian, Idaho
  - EndoCeutics site # 27, Baltimore, Maryland
  - EndoCeutics site # 22, Kalamazoo, Michigan
  - EndoCeutics site # 25, Lincoln, Nebraska
  - EndoCeutics site # 28, Moorestown, New Jersey
  - EndoCeutics site # 44, New Brunswick, New Jersey
  - EndoCeutics site # 19, New York, New York
  - EndoCeutics site # 16, Durham, North Carolina
  - EndoCeutics site # 05, Cleveland, Ohio
  - EndoCeutics site # 15, Columbus, Ohio
  - EndoCeutics site # 35, Pittsburgh, Pennsylvania
  - EndoCeutics site # 09, West Jordan, Utah
  - EndoCeutics site # 31, Charlottesville, Virginia
  - EndoCeutics site # 03, Norfolk, Virginia
- Canada (9):
  - EndoCeutics site # 13, Calgary, Alberta
  - EndoCeutics site # 06, Bathurst, New Brunswick
  - EndoCeutics site # 04, Drummondville, Quebec
  - EndoCeutics site # 12, Montreal, Quebec
  - EndoCeutics site # 02, Québec, Quebec
  - EndoCeutics site # 01, Québec, Quebec
  - EndoCeutics site # 18, Saint Romuald, Quebec
  - EndoCeutics site # 08, Shawinigan, Quebec
  - EndoCeutics site # 11, Sherbrooke, Quebec

REFERENCES:
- [Result] Archer DF, Labrie F, Bouchard C, Portman DJ, Koltun W, Cusan L, Labrie C, Cote I, Lavoie L, Martel C, Balser J; VVA Prasterone Group. Treatment of pain at sexual activity (dyspareunia) with intravaginal dehydroepiandrosterone (prasterone). Menopause. 2015 Sep;22(9):950-63. doi: 10.1097/GME.0000000000000428. PMID 25734980
- [Result] Portman DJ, Labrie F, Archer DF, Bouchard C, Cusan L, Girard G, Ayotte N, Koltun W, Blouin F, Young D, Wade A, Martel C, Dube R; other participating members of VVA Prasterone Group. Lack of effect of intravaginal dehydroepiandrosterone (DHEA, prasterone) on the endometrium in postmenopausal women. Menopause. 2015 Dec;22(12):1289-95. doi: 10.1097/GME.0000000000000470. PMID 25968836
- [Result] Martel C, Labrie F, Archer DF, Ke Y, Gonthier R, Simard JN, Lavoie L, Vaillancourt M, Montesino M, Balser J, Moyneur E; other participating members of the Prasterone Clinical Research Group. Serum steroid concentrations remain within normal postmenopausal values in women receiving daily 6.5mg intravaginal prasterone for 12 weeks. J Steroid Biochem Mol Biol. 2016 May;159:142-53. doi: 10.1016/j.jsbmb.2016.03.016. Epub 2016 Mar 10. PMID 26972555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 464 subjects were screened at 33 medical/research sites located in the US (24 centers) and Canada (9 centers) and 255 subjects were randomized. The first subject first visit was on 30-NOV-2010 and the last subject last visit was on 29-JUL-2011.
Groups:
- 0.50% DHEA: DHEA: Vaginal suppository containing 0.50% (6.5 mg) DHEA; daily dosing with one suppository for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Started | 81 | 87 | 87
Safety Population | 80 | 86 | 87
ITT Population | 77 | 79 | 81
Completed | 72 | 74 | 76
Not Completed | 9 | 13 | 11
Not completed — Adverse Event | 1 | 4 | 2
Not completed — Withdrawal by Subject | 4 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Entry criteria not met/non-compliance | 4 | 7 | 6

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population corresponds to the Safety Population which includes all subjects who received any amount of DHEA or placebo, and who have any safety information available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | Total
Number analyzed (Participants) | 80 | 86 | 87 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.81 (5.89) | 59.37 (6.39) | 57.51 (5.63) | 58.55 (6.01)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 80 | 86 | 87 | 253
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Caucasian | 69 | 81 | 83 | 233
  Black or African American | 9 | 4 | 3 | 16
  Asian | 1 | 0 | 1 | 2
  Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Percentage of Parabasal Cells in the Maturation Index of the Vaginal Smear
Description: The percentage of parabasal cell was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including the basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: Efficacy analyses were performed primarily on the Intent to Treat (ITT) population defined as all subjects who have received at least one dose of study drug with a baseline (Day 1) evaluation meeting the study entry criteria.
Measure: Mean (Standard Error); unit: Percentage of parabasal cells
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 77 | 79 | 81
Percentage of parabasal cells
  Baseline | 68.48 (4.41) | 65.72 (4.56) | 65.05 (4.63)
  Week 12 | 66.86 (4.37) | 28.43 (3.62) | 17.65 (2.87)
  Change from Baseline to Week 12 | -1.62 (3.22) | -37.29 (4.16) | -47.40 (4.72)

2. Primary Outcome: Change From Baseline to Week 12 in Percentage of Superficial Cells in the Maturation Index of the Vaginal Smear
Description: The percentage of superficial cell was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including the basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: Efficacy analyses were performed primarily on the Intent-to-Treat (ITT) population defined as all subjects who have received at least one dose of study drug with a baseline (Day 1) evaluation meeting the study entry criteria.
Measure: Mean (Standard Error); unit: Percentage of superficial cells
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 77 | 79 | 81
Percentage of superficial cells
  Baseline | 0.73 (0.15) | 0.68 (0.13) | 0.68 (0.12)
  Week 12 | 1.64 (0.33) | 5.43 (0.57) | 6.30 (0.59)
  Change from Baseline to Week 12 | 0.91 (0.31) | 4.75 (0.58) | 5.62 (0.61)

3. Primary Outcome: Change From Baseline to Week 12 in Vaginal pH
Description: A pH strip fixed on an Ayre spatula (or equivalent) was applied directly to the lateral wall of the vagina. The change in color of the pH indicator strip was compared to the color chart for pH evaluation. The corresponding pH value (with one decimal) was recorded. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 77 | 79 | 81
units on a scale
  Baseline | 6.51 (0.07) | 6.48 (0.07) | 6.47 (0.07)
  Week 12 | 6.31 (0.09) | 5.70 (0.11) | 5.43 (0.10)
  Change from Baseline to Week 12 | -0.21 (0.08) | -0.77 (0.10) | -1.04 (0.11)

4. Primary Outcome: Change From Baseline to Week 12 in Severity of the Most Bothersome Symptom of Dyspareunia
Description: The severity of dyspareunia was evaluated by a questionnaire filled out by women. The severity of dyspareunia recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 77 | 79 | 81
units on a scale
  Baseline | 2.58 (0.06) | 2.56 (0.06) | 2.63 (0.05)
  Week 12 | 1.71 (0.11) | 1.54 (0.12) | 1.36 (0.12)
  Change from Baseline to Week 12 | -0.87 (0.11) | -1.01 (0.11) | -1.27 (0.11)

5. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Dryness
Description: The severity of vaginal dryness was evaluated by a questionnaire filled out by women. The severity of vaginal dryness recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: Efficacy analyses on vaginal dryness were performed on a sub-group of the Intent to Treat (ITT) population (defined as all subjects who have received at least one dose of study drug with a baseline (Day 1) evaluation meeting the study entry criteria) who have self-identified moderate to severe vaginal dryness at Baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 60 | 70 | 62
units on a scale
  Baseline | 2.33 (0.06) | 2.20 (0.05) | 2.37 (0.06)
  Week 12 | 1.32 (0.12) | 0.91 (0.10) | 0.92 (0.10)
  Change from Baseline to Week 12 | -1.02 (0.14) | -1.29 (0.11) | -1.45 (0.12)

6. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Secretions
Description: To evaluate the aspect of the mucosa and the local tolerance to DHEA suppositories, the vaginal secretions (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy were then analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: Analyses were performed primarily on the Intent to Treat (ITT) population defined as all subjects who have received at least one dose of study drug with a baseline (Day 1) evaluation meeting the study entry criteria.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 77 | 79 | 81
units on a scale
  Baseline | 2.78 (0.08) | 2.81 (0.07) | 2.83 (0.08)
  Week 12 | 2.36 (0.08) | 2.10 (0.09) | 1.95 (0.08)
  Change from Baseline to Week 12 | -0.42 (0.08) | -0.71 (0.09) | -0.88 (0.11)

7. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Epithelial Integrity
Description: To evaluate the aspect of the mucosa and the local tolerance to DHEA suppositories, the vaginal epithelial integrity (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was then analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 77 | 79 | 81
units on a scale
  Baseline | 2.58 (0.09) | 2.57 (0.10) | 2.57 (0.10)
  Week 12 | 2.13 (0.09) | 1.92 (0.09) | 1.69 (0.09)
  Change from Baseline to Week 12 | -0.45 (0.08) | -0.65 (0.09) | -0.88 (0.10)

8. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Epithelial Surface Thickness
Description: To evaluate the aspect of the mucosa and the local tolerance to DHEA suppositories, the vaginal epithelial surface thickness (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was then analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 77 | 79 | 81
units on a scale
  Baseline | 2.91 (0.07) | 2.90 (0.08) | 2.89 (0.07)
  Week 12 | 2.57 (0.08) | 2.32 (0.09) | 2.14 (0.08)
  Change from Baseline to Week 12 | -0.34 (0.07) | -0.58 (0.09) | -0.75 (0.09)

9. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Color
Description: To evaluate the aspect of the mucosa and the local tolerance to DHEA suppositories, the vaginal color (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was then analyzed using the values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 77 | 79 | 81
units on a scale
  Baseline | 2.82 (0.08) | 2.94 (0.08) | 2.94 (0.08)
  Week 12 | 2.56 (0.08) | 2.27 (0.10) | 2.05 (0.09)
  Change from Baseline to Week 12 | -0.26 (0.07) | -0.67 (0.09) | -0.89 (0.10)

ADVERSE EVENTS:
Time Frame: From Baseline up to 12 Weeks (+ 30-day follow-up period after last dose)
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Serious Adverse Events (participants affected / at risk) | 0/80 | 3/86 | 1/87
Other Adverse Events (participants affected / at risk) | 9/80 | 12/86 | 10/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | 0.25% DHEA (N=86) | 0.50% DHEA (N=87)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Bone abscess (Infections and infestations) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | 0.25% DHEA (N=86) | 0.50% DHEA (N=87)
Application site discharge (General disorders) | 5 | 6 | 5
Urinary tract infection (Infections and infestations) | 4 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall provide to the SPONSOR 30 days prior to submission all documents for publication, presentation, etc that report any trial results. The SPONSOR shall have editorial rights on documents and the right to review/comment with regard to (1) proprietary information, (2) accuracy of the information, (3) correctness of the scientific evaluation/conclusions and (4) to ensure that the information is fairly balanced and in compliance with regulations.